CLINICAL TRIAL: NCT00737373
Title: A Multicenter, Randomised Phase II Trial on the Therapy of Advanced Gastric Cancer or Adenocarcinoma of the Esophagogastric Junction in Patients Older Than 65 Years With Specific Regard of Quality of Life and Pharmacogenetic Risk Profile
Brief Title: Oxaliplatin and 5-Fluorouracil With or Without Docetaxel in Elderly Patients (>65 y) With Stomach and Esophagus Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLOT65+
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-08

CONDITIONS: Gastric Cancer; Adenocarcinoma of the Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): FLOT
  Interventions: Drug: Docetaxel; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: folinic acid
- 2 (Active Comparator): FLO
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: folinic acid

INTERVENTIONS:
Drug: Docetaxel — 50mg/m2 qd15
  Arms: 1
Drug: 5-Fluorouracil — 2600mg/m2 qd15
Drug: Oxaliplatin — 85mg/m2 qd15
Drug: folinic acid — 200mg/m2 qd15

SUMMARY:
In this trial, FLOT will be evaluated as therapy option for elderly patients (>65 years) with advanced gastric cancer in comparison to the well established FLO scheme. The hypothesis is that FLOT is more effective than FLO in elderly patients with acceptable side effects.

DETAILED DESCRIPTION:
Patients with locally advanced, potentially operable or metastatic gastric cancer or adenocarcinoma of the esophagogastric junction without prior therapy in the palliative setting are treated with:

* Arm A: FLO
* Arm B: FLOT

max. 12 cycles

Evaluation of quality of life by standard forms at baseline and then every 2 months until progress of disease. Pharmacogenetic analyses will be done to evaluate a risk profile for platin-based therapies. 140 patients will be treated (70 per arm)

primary endpoint:

* Response Rate

secondary endpoints:

* Prospective Validation of a pharmacogenetic risk profile for patients with advanced GC under first-line therapy with platin/docetaxel
* Evaluation of quality of life
* safety and tolerability
* progression free survival (PFS), time to treatment failure (TTF), overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* metastatic or locally advanced gastric cancer or adenocarcinoma of the esophagogastric junction
* no prior chemotherapy in metastatic state
* adequate blood and biochemistry parameters

Exclusion Criteria:

* hypersensitivity for 5-FU, Leucovorin, Oxaliplatin or Docetaxel
* KHK, cardiomyopathy or cardiac insufficiency
* malignancy <5 years ago
* brain metastases
* severe internal disease or inadequate blood and biochemistry parameters

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 143 (Actual)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
response (WHO criteria) | staging every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, MD, Study Chair — Krankenhaus Nordwest
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

REFERENCES:
- [Background] Al-Batran SE, Hartmann JT, Probst S, Schmalenberg H, Hollerbach S, Hofheinz R, Rethwisch V, Seipelt G, Homann N, Wilhelm G, Schuch G, Stoehlmacher J, Derigs HG, Hegewisch-Becker S, Grossmann J, Pauligk C, Atmaca A, Bokemeyer C, Knuth A, Jager E; Arbeitsgemeinschaft Internistische Onkologie. Phase III trial in metastatic gastroesophageal adenocarcinoma with fluorouracil, leucovorin plus either oxaliplatin or cisplatin: a study of the Arbeitsgemeinschaft Internistische Onkologie. J Clin Oncol. 2008 Mar 20;26(9):1435-42. doi: 10.1200/JCO.2007.13.9378. PMID 18349393
- [Background] Al-Batran SE, Hartmann JT, Hofheinz R, Homann N, Rethwisch V, Probst S, Stoehlmacher J, Clemens MR, Mahlberg R, Fritz M, Seipelt G, Sievert M, Pauligk C, Atmaca A, Jager E. Biweekly fluorouracil, leucovorin, oxaliplatin, and docetaxel (FLOT) for patients with metastatic adenocarcinoma of the stomach or esophagogastric junction: a phase II trial of the Arbeitsgemeinschaft Internistische Onkologie. Ann Oncol. 2008 Nov;19(11):1882-7. doi: 10.1093/annonc/mdn403. Epub 2008 Jul 31. PMID 18669868
- [Background] Al-Batran SE, Atmaca A, Hegewisch-Becker S, Jaeger D, Hahnfeld S, Rummel MJ, Seipelt G, Rost A, Orth J, Knuth A, Jaeger E. Phase II trial of biweekly infusional fluorouracil, folinic acid, and oxaliplatin in patients with advanced gastric cancer. J Clin Oncol. 2004 Feb 15;22(4):658-63. doi: 10.1200/JCO.2004.07.042. PMID 14966088
- [Derived] Al-Batran SE, Pauligk C, Homann N, Hartmann JT, Moehler M, Probst S, Rethwisch V, Stoehlmacher-Williams J, Prasnikar N, Hollerbach S, Bokemeyer C, Mahlberg R, Hofheinz RD, Luley K, Kullmann F, Jager E. The feasibility of triple-drug chemotherapy combination in older adult patients with oesophagogastric cancer: a randomised trial of the Arbeitsgemeinschaft Internistische Onkologie (FLOT65+). Eur J Cancer. 2013 Mar;49(4):835-42. doi: 10.1016/j.ejca.2012.09.025. Epub 2012 Oct 11. PMID 23063354